CLINICAL TRIAL: NCT01509521
Title: The Oxygenation of the Brain During Caesarean Section. A Comparison of Ephedrine Versus Phenylephrine
Brief Title: The Oxygenation of the Brain During Caesarean Section
Acronym: OBDUC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Naestved Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Visti Foss, Principal Investigator, Naestved Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-006103-35; SJ-271 (Other: Sponsor´s protocol code number)
Record Dates: First submitted 2012-01-08; First posted 2012-01-13 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Complications; Cesarean Section
Keywords: Spectroscopy, Near-Infrared; Fetal heartrate; Ephedrine; Phenylephrine
MeSH Terms: interventions — Ephedrine; Phenylephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ephedrine (Active Comparator)
  Interventions: Drug: Ephedrine
- Phenylephrine (Active Comparator)
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Ephedrine — An infusion with a maximum of 3 mg/minute for maximum 60 minutes or if sideeffects develope.
  Other Names: Efedrin; Ephedrine hydrochloride
  Arms: Ephedrine
Drug: Phenylephrine — An infusion of maximum 4 mg/hour for maximum 60 minutes.
  Other Names: Phenylephrine Hydrochloride; Metaoxedrin
  Arms: Phenylephrine

SUMMARY:
The purpose of this study is to determine the impact of phenylephrine versus ephedrine on organ perfusion, in women undergoing caesarean section receiving spinal anaesthesia. The organ perfusion is estimated by measuring the maternal cerebral oxygenation by NIRS(Near-infrared spectroscopy)and the foetal heartrate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women
* Over 18 years old
* ASA 1-2
* Undergoing elective caesarean section
* Height over 160 cm or under 180 cm

Exclusion Criteria:

* Allergic reactions to ephedrine or phenylephrine
* High blood levels of bilirubin
* HELPP syndrome
* Preeclampsia (pregnancy-induced hypertension)
* Non singleton pregnancies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Frontal lobe cerebral oxygenation | Participants will be followed for the time in the operation theatre of the hospital stay, an expected average of 1 hour
  Determine the frontal lobe cerebral oxygantion by Near-Infrared Spectroscopy (NIRS),from before induction of spinal anaesthesia to end of surgery.
Foetal heartrate | Participants will be followed for the time in the operation theatre of the hospital stay, an expected average of 1 hour
  From before induction of spinal anaesthesia to 15 min after delivery

SECONDARY OUTCOMES:
Mean arterial pressure | Participants will be followed for the time in the operation theatre of the hospital stay, an expected average of 1 hour
  The mean arterial pressure is measures from before induction of spinal anaesthesia to end of surgery.
Cardiac output | Participants will be followed for the time in the operation theatre of the hospital stay, an expected average of 1 hour
  The cardiac output is measures from before induction of spinal anaesthesia to end of surgery.
Umbilical cord pH and Base excess | Blood analysis taken immediately after the the clamping of the umbilical cord, an average of 20 minutes.
  The umbilical cord blood analysis for evaluation of the newborn's acid-base status is taken immediately after delivery. It is the most objective way of assessing the fetal metabolic condition at birth.

CONTACTS AND LOCATIONS:
Overall Officials: Visti Foss, Principal Investigator — Naestved Hospital
Locations (1):
- Naestved Hospital, Næstved, Denmark

REFERENCES:
- [Derived] Chooi C, Cox JJ, Lumb RS, Middleton P, Chemali M, Emmett RS, Simmons SW, Cyna AM. Techniques for preventing hypotension during spinal anaesthesia for caesarean section. Cochrane Database Syst Rev. 2020 Jul 1;7(7):CD002251. doi: 10.1002/14651858.CD002251.pub4. PMID 32619039
- [Derived] Foss VT, Christensen R, Rokamp KZ, Nissen P, Secher NH, Nielsen HB. Effect of phenylephrine vs. ephedrine on frontal lobe oxygenation during caesarean section with spinal anesthesia: an open label randomized controlled trial. Front Physiol. 2014 Mar 3;5:81. doi: 10.3389/fphys.2014.00081. eCollection 2014. PMID 24624090